CLINICAL TRIAL: NCT03446820
Title: Sleep Quality and Microclimate Study
Brief Title: This Study Assesses the Impact of Different Sheets on Body Temperature and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 18-000832
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to sleep in the residential module of the Well Living Lab. One week will be with standard sheets, followed by one week of hygro cotton sheets.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep participants (Other): Crossover from standard sheets to hygro cotton sheets
  Interventions: Other: hygro cotton sheets

INTERVENTIONS:
Other: hygro cotton sheets — hygro cotton sheets will be utilized to impact microclimate

SUMMARY:
Thermal comfort and subsequent sleep quality will improve with the use of bedding that incorporates thermoregulation technology, in comparison to standard bedding products.

DETAILED DESCRIPTION:
Participants will spend nights sleeping in the residential module of the Well Living Lab. Participants will cross over from normal sheets to hygro cotton sheets to assess impact of different sheet types on microclimate (e.g. temperature) and the impact on sleep quality.

ELIGIBILITY:
Inclusion Criteria. Premenopausal women Age 21-45

Exclusion Criteria History of sleep disorders

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal women
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
body temperature | 1 night
  body temperature collected via body sensors

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Bauer, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota